CLINICAL TRIAL: NCT00572078
Title: Phase I Dose-Escalation Drug-Interaction Study of Sorafenib and Bevacizumab in Combination With Paclitaxel in Patients With Solid Tumors
Brief Title: Sorafenib and Bevacizumab in Combination With Paclitaxel in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Safi Shahda (Other)
Collaborators: Genentech, Inc. (Industry); Bayer (Industry)
Responsible Party: Sponsor-Investigator, Safi Shahda, Principal Investigator, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0706-05 IUCRO-0171
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: SOLID TUMORS
Keywords: solid tumor
MeSH Terms: interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib, Bevacizumab & Paclitaxel (Experimental): Paclitaxel is given as i.v infusion over 60 min on days 1, 8, 15 every 28 days. Sorafenib is given orally starting with cycle 1 day 2. Bevacizumab is given as i.v infusion on days 1 and 15 every 28 days.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Cohort 1 200 mg po BID D1-5; Cohort 2 200 mg po BID; Cohort 3 400 mg po BID D1-5 Cohort 4 400 mg po BID
  Other Names: Bay 43-9006

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability and describe the maximum tolerated dose (MTD) of treatment with escalating doses of sorafenib in combination with bevacizumab and paclitaxel for patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of a solid tumor with evidence of residual, recurrent, or metastatic disease. Patients must be incurable by surgical or other standard available therapy
* Measurable or evaluable disease; tumor size of ≥ 2 cm on CT scan
* Patients may have received prior standard taxane therapy or anti-VEGF therapy, but may not have progressed on both therapies. Progression on one type therapy (either taxane or anti-VEGF) is allowed

Exclusion Criteria:

* History or presence of central nervous system (CNS) disease (i.e., primary brain tumor, malignant seizures, CNS metastases or carcinomatous meningitis).
* Prior chemotherapy ≤ 3 weeks prior to registration. Patients must have recovered from all therapy-related toxicities
* Prior biologic or immunotherapy ≤ 3 weeks prior to registration. Patients must have recovered from all therapy-related toxicities
* Prior full pelvic field radiotherapy ≤ 4 weeks or limited field radiotherapy ≤ 2 weeks prior to randomization. Patients must have recovered to less than or equal to grade 1 from all therapy-related toxicities except alopecia. The site of previous radiotherapy should have evidence of progressive disease if this is the only site of evaluable disease
* Major surgery (i.e., laparotomy) ≤ 4 weeks prior to randomization or anticipation of need for major surgical procedure during the course of the study
* Minor surgery ≤ 2 weeks prior to randomization. Insertion of a vascular access device is not considered major or minor surgery in this regard. Patients must have recovered from all surgery-related toxicities
* Peripheral neuropathy with functional impairment ≥ Common Terminology Criteria (CTC) grade 2 neuropathy, regardless of causality
* Pleural effusion or ascites that causes respiratory compromise (≥ CTC grade 2 dyspnea)
* Concurrent severe and/or uncontrolled cardiac, vascular or infectious conditions (as described in the protocol) which could compromise participation in the study
* Patients at risk of QT prolongation such as patients with congenital long QT syndrome or with long corrected QT (QTc) at baseline (i.e. QTc greater than 450 msec in males, and greater than 470 msec in females) will be excluded
* Lung carcinoma of squamous cell histology (mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible; sputum cytology alone is not acceptable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-01-23 (Actual); Primary Completion 2011-01-04 (Actual); Study Completion 2014-09-14 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability and describe the maximum tolerated dose (MTD) of treatment with escalating doses of sorafenib in combination with bevacizumab and paclitaxel for patients with advanced solid tumors. | baseline through end of treatment

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of paclitaxel and sorafenib alone and in combination | baseline through end of treatment
To evaluate pharmacodynamic changes a)in tumor vascular parameters and b)in plasma VEGF and soluble VEGF receptor levels, and correlate with clinical outcomes and sorafenib pharmacokinetic (PK) profile. | baseline through end of treatment
To evaluate variants in genes of paclitaxel drug-metabolism and drug-transporters P glycoprotein and correlate with PK profile for paclitaxel and with clinical outcomes | baseline through end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Safi G Shahda, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Chiorean EG, Perkins SM, Strother RM, Younger A, Funke JM, Shahda SG, Hahn NM, Sandrasegaran K, Jones DR, Skaar TC, Schneider BP, Sweeney CJ, Matei DE. Phase I, Pharmacogenomic, Drug Interaction Study of Sorafenib and Bevacizumab in Combination with Paclitaxel in Patients with Advanced Refractory Solid Tumors. Mol Cancer Ther. 2020 Oct;19(10):2155-2162. doi: 10.1158/1535-7163.MCT-20-0277. Epub 2020 Aug 26. PMID 32847973